CLINICAL TRIAL: NCT04484896
Title: Effects of Message Framing on Recruiting Rh-D Negative Blood Donors in an Emergency Situation
Brief Title: Message Framing on Recruiting Rh-D Negative Blood Donors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Blood Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Recruiting Rh-D- blood donors
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Blood Donation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant did not know the difference between the three message.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gain-frame Message (Experimental): Short messaging service (SMS) message: Dear group O/A Rh-D negative blood donor:
  Hello! The inventory of group O/A Rh-D negative blood product is low at present, but patients with such blood group are in urgent need of blood. If you can, please consider donating blood again to save lives. Thank you for your support.
  Please bring your identification (ID) card and show this message to our staff. Thank you.
  Interventions: Other: Gain-framed SMS message
- Loss-frame Message (Experimental): SMS message: Dear group O/A Rh-D negative blood donor:
  Hello! The inventory of group O/A Rh-D negative blood product is low at present, but patients with such blood group are in urgent need of blood. If you can, please consider donating blood again to prevent the loss of life. Thank you for your support.
  Please bring your ID card and show this message to our staff. Thank you.
  Interventions: Other: Loss-framed SMS message
- Information Message (Experimental): SMS message: Dear group O/A Rh-D negative blood donor:
  Hello! The inventory of group O/A Rh-D negative blood product is low at present, if you can, please consider donating blood again. Thank you for your support.
  Please bring your ID card and show this message to our staff. Thank you.
  Interventions: Other: Information SMS message
- Control group (No Intervention): Donors in this group were not received SMS reminders.

INTERVENTIONS:
Other: Gain-framed SMS message — Emergency recruitment cell phone short messages that emphasizing donating blood can save patients' lives were sent to donors in this group.
  Arms: Gain-frame Message
Other: Loss-framed SMS message — Emergency recruitment cell phone short messages emphasizing that donating blood can prevent patients from death were sent to donors in this group.
  Arms: Loss-frame Message
Other: Information SMS message — Emergency recruitment cell phone short messages that only mentioning the low Rh-negative blood stockpile were sent to donors in this group.
  Arms: Information Message

SUMMARY:
Rh negative blood group is a rare blood group in China, as it only accounts for 0.3-0.4 percent of the Han population. Therefore, low inventory is often found in blood collection and supply agencies in many regions in China. On July 22, 2020 blood stockpile of O-negative and A-negative in Guangzhou Blood Center reached the warning line, and we took measures for emergency recruitment. O-negative and A-negative blood donors whose last donation dates were between January 1, 2018 and December 31, 2019 were identified and randomly assigned to four groups. Three different recruitment text messages were send three groups. We observed the re-donation rates among four groups within one week.

ELIGIBILITY:
Inclusion Criteria:

- O and A Rh- negative blood donors Last donations were between January 1, 2018 and December 31, 2019

Exclusion Criteria:

- With an obviously invalid phone number Serological results of the last donation were positive

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1082 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2020-07-29 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Re-donation rate | 7 days
  Intention-to-treat were applied. Re-donation rate was defined as the number of donors in each group divided by donors who re-donated within 7 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Blood Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided